CLINICAL TRIAL: NCT05024136
Title: Study on the Efficacy of Vetiver Essential Oil Aroma on Depression/Anxiety People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, Associate Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CS1-20030
Record Dates: First submitted 2021-05-20; First posted 2021-08-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Anxiety Depression Disorder
Keywords: Vetiver oil; Aromatherapy; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Subjects take 30 mins aromatherapy of Limon essential oil per time, a total of 3 times for the month.
  Interventions: Device: Limon essential oil aromatherapy
- Experimental (Experimental): Subjects take 30 mins aromatherapy of vetiver essential oil per time, a total of 3 times for the month.
  Interventions: Device: Vetiver essential oil aromatherapy

INTERVENTIONS:
Device: Limon essential oil aromatherapy — Subjects receive three times 30 mins aromatherapy of Limon essential oil per time for the month. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), autonomic nerve parameters including a. SDNN (standard deviation of all normal to normal intervals index); b. HRV（heart rate variability）; c. LF（0.04-0.15 Hz）and HF（0.15-0.4 Hz）were measured every week. PSQI（Pittsburgh sleep quality index）and HADS (Hospital Anxiety and Depression Scale) were measured initial and ten ends.
  Arms: Placebo
Device: Vetiver essential oil aromatherapy — Subjects receive three times 30 mins aromatherapy of vetiver essential oil per time for the month. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), autonomic nerve parameters including a. SDNN (standard deviation of all normal to normal intervals index); b. HRV（heart rate variability）; c. LF（0.04-0.15 Hz）and HF（0.15-0.4 Hz）were measured every week. PSQI（Pittsburgh sleep quality index）and HADS (Hospital Anxiety and Depression Scale) were measured initial and ten ends.
  Arms: Experimental

SUMMARY:
In this study, subjects with depression/anxiety inhaled the essential oil, which contained sedative, soothing, and relaxing active ingredients to stimulate the olfactory nerve. The essential oil further transmitted to the limbic system that controls emotions in the brain, and then affected the human's mood. The natural aroma can not only awaken the limbic system's memory of aroma but also reflect the subconscious area of the brain, with physiological changes (such as controlling blood pressure, breathing, heartbeat, stress changes, memory, and hormonal coordination.) This study monitors the subject's autonomic nerve parameters before and after aromatherapy to obtain the olfactory cerebral nervous system to convey the message. When the study finishes, we expected to help the subject to relax and soothe the mind.

DETAILED DESCRIPTION:
Subjects receive three times 30 mins aromatherapy of Limon or Vetiver essential oil per time for the month. Anthropometric measurements such as blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), autonomic nerve parameters including a. SDNN (standard deviation of all normal to normal intervals index); b. HRV（heart rate variability）; c. LF（0.04-0.15 Hz）and HF（0.15-0.4 Hz）were measured every week. PSQI（Pittsburgh sleep quality index）and HADS (Hospital Anxiety and Depression Scale) were measured initial and ten ends.

ELIGIBILITY:
Inclusion Criteria:

1. Depressed/anxious people (diagnosed as a single episode of major depression, recurrence of major depression, mild depression, panic disorder, and anxiety.) Those diagnosed with symptoms of depression, and anxiety related to stress adjustment disorder, and willing to cooperate with the study.
2. Age 20-65 years old

Exclusion Criteria:

1. an alcoholic
2. Uncontrolled diabetes
3. Those who have had a stroke in the last year
4. Pregnant and lactating women
5. People with liver or heart disease
6. Arrhythmia or those with a heart rhythm regulator
7. Those whose heart has already been fitted with a cardiac catheter stent
8. Those who have used central nervous system stimulants (regardless of the length of time)
9. Those who are allergic to essential oils
10. Those who have used aromatherapy within a month
11. Subjects request to withdraw from the trial
12. The host feels unsuitable to continue the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The aromatherapy measure autonomic nerve parameter SDNN (standard deviation of all normal to normal intervals index) | one month
The measure blood pressure (SBP and DBP) | one month
  values change of systolic and diastolic BPs

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan